CLINICAL TRIAL: NCT05134922
Title: Expanded Access Protocol for Subjects Previously Treated With Gedatolisib in a Celcuity-Sponsored Clinical Study (B2151009)
Brief Title: Expanded Access Protocol for Subjects Previously Treated With Gedatolisib in B2151009
Status: Available | Type: Expanded Access
Sponsor: Celcuity Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CELC-G-001
Record Dates: First submitted 2021-11-14; First posted 2021-11-26 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Breast Neoplasm Malignant Female
MeSH Terms: interventions — gedatolisib

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Gedatolisib — Gedatolisib is a potent, reversible dual inhibitor that selectively targets phosphoinositide 3 kinase (PI3K) and mammalian target of rapamycin (mTOR) in biochemical and cellular assays.

SUMMARY:
Continued access to treatment for subjects who continue benefit from therapy with gedatolisib in combination with palbociclib, and fulvestrant or letrozole.

DETAILED DESCRIPTION:
The primary purpose of this study is to provide continuing access to treatment for subjects who continue benefit from therapy with gedatolisib in combination with palbociclib, and fulvestrant or letrozole.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled in the B2151009 clinical study and benefiting from treatment with gedatolisib in combination with other therapies as determined by the Investigator
2. Previously demonstrated compliance and are willing and able to comply with scheduled visits, treatment plans, and other study procedures
3. No evidence of progressive disease, as determined by the Investigator
4. Provide written informed consent prior to enrolling and receiving treatment

Exclusion Criteria:

1. Permanently discontinued from treatment in Study B2151009, or discontinued from Study B2151009 for any reason
2. Women who are pregnant, intend to become pregnant, or nursing

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Michigan, Ann Arbor, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington